CLINICAL TRIAL: NCT00518635
Title: Effects of Low Dose Growth Hormone (GH) Therapy on Insulin Sensitivity, Metabolic Profile, Adipocyte IGF-I and Insulin Signaling, Intramyocellular Lipids, and Cortisol Metabolism in Obese Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Low Dose Growth Hormone in Obese PCOS Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kevin Yuen, Associate Professor in Endocrinology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB3711
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Growth hormone; Insulin sensitivity; Polycystic ovary
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Human Growth Hormone; Growth Hormone; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Growth hormone or Placebo 0.1 mg/day self-administrated once a day.
  Interventions: Drug: Nutropin

INTERVENTIONS:
Drug: Nutropin — Nutropin 0.1 mg/day self-administered once a day
  Other Names: Growth hormone, PCOS, insulin sensitivity

SUMMARY:
Study hypothesis:

Growth hormone (GH), through its generation of free 'bioavailable' insulin-like growth factor (IGF)-I, can improve insulin sensitivity and the metabolic profile of women with polycystic ovary syndrome.

Study aims:

To determine the mechanism of how low dose GH treatment affects the body's sensitivity to insulin actions and whether this low GH dose can affect the body's handling of steroid hormone levels (cortisol clearance) and testosterone (male hormones) in obese women with polycystic ovary syndrome.

Study design:

Obese women with polycystic ovary syndrome, but not recently been on GH treatment, and presently attending Outpatients Clinic will be invited to participate in this study. The subjects will be assessed at the initial visit to ascertain their suitability before further participating in the study. If suitable, an equal number of women will be randomized to receive either daily low dose GH or placebo injections first for 12 weeks, before exchanging over for another 12 weeks of treatment after a 4-week washout period. Before, during and after treatment, the subjects will be assessed at frequently with blood tests, scans and fat biopsies. During the study, the subjects will be studied 4 times at the Oregon Clinical and Translational Research Institute (OCTRI). At the first, second and final visit, testing will include scans to measure the amount of whole body fat and fat in the stomach area, muscle, and liver; blood tests to measure levels of cortisol, and fat tissue (taken from a biopsy) analysis to measure the density of insulin-like growth factor-I (a hormone stimulated by growth hormone in the body) in fat; whereas blood tests to examine how well insulin works in the body (insulin sensitivity) will be collected at all visits of the study.

DETAILED DESCRIPTION:
The study will be a double-blinded cross-over study. Thirty subjects will be screened for eligibility initially, and the first 12 eligible subjects will be enrolled. Six subjects will be randomized to receive the low GH dose (0.1 mg/day) treatment and 6 subjects to receive Placebo treatment for 12 weeks, exchanging their treatment for a further 12 weeks after a 4-week washout period. The study drugs will be stored at the Oregon Health and Science University (OHSU) Research Pharmacy and following randomization, the subjects will be taught by our Endocrine Nurses to self-administer the subcutaneous GH and Placebo injections using Nutropin/Placebo vials and insulin syringes into the abdomen at 2200h. Randomization for treatment assignment will be performed by an investigator not directly involved in the patients' recruitment, treatment and follow-up care. The randomization process will be performed by computerized pre-assigned random codes by blocks, stratified by age and examined for possible differences in body mass index. During their in-patient stay at the Oregon Clinical and Translational Research Institute (OCTRI) at OHSU, subjects will only be allowed to eat the food provided to them by the OCTRI.

Initial Screening Assessment (outpatient)

The following assessments will be performed:

* Written informed consent
* Demographics (demographic information including the subject's birth date, and race)
* Physical exam and medical history
* Previous/significant medical history
* Concomitant medication review
* Vital signs, e.g., pulse and blood pressure measurements
* Height and weight
* Laboratory findings, e.g. CBC, electrolytes, and fasting glucose levels

  * Visit 1, Baseline Assessment for the First Treatment Phase (in-patient)

The following is a description of the assessments that will be performed after consent is obtained:

* Physical exam and medical history
* Vital signs, e.g., pulse and blood pressure measurements
* Height and weight
* Waist circumference measurement
* Concomitant medication review
* Urine pregnancy test
* Fasting blood assessments, e.g., hemoglobin, glucose, insulin, C-peptide, serum total and free IGF-I, IGFBP-3, C-reactive protein, non-esterified fatty acids (NEFAs), testosterone, albumin, sex hormone binding globulin and androstenedione
* A 3-hour one-step hyperinsulinemic euglycemic clamp
* MRS and DEXA scans
* Cortisol clearance rate assessments
* Fat biopsy
* Randomization to GH or Placebo
* Teach GH or Placebo self-administration

  * Visit 2, Final Assessment for the First Treatment Phase (Week 12 +/- 1 week) (outpatient)

The following is a description of the assessments that will be performed at the end of the first treatment phase with either GH or Placebo. Subjects will also be monitored for safety with the collection of the following:

* Physical exam and medical history
* Vital signs, e.g. pulse and blood pressure measurements
* Height and weight
* Waist circumference measurement
* Concomitant medication review
* Adverse event recording
* Urine pregnancy test
* Fasting blood assessments, e.g. hemoglobin, glucose, insulin, C-peptide, serum total and free IGF-I, IGFBP-3, C-reactive protein, adiponectin, ghrelin, non-esterified fatty acids (NEFAs), testosterone, albumin, sex hormone binding globulin and androstenedione
* A 3-hour one-step hyperinsulinemic euglycemic clamp
* MRS and DEXA scans
* Cortisol clearance rate assessments
* Fat biopsy

Washout Period and Crossover After the first treatment phase with GH or Placebo, the subjects will have a 4-week washout period and the treatment will be crossed over for another 12-week treatment phase with either GH or Placebo. During this time, the subjects will be advised to maintain a stable diet and weight.

Visit 3, Baseline Assessment for the Second Treatment Phase (Week 16 +/- 1 week) (as outpatient)

The following is a description of the assessments that will be performed:

* Physical exam and medical history
* Vital signs, e.g., pulse and blood pressure measurements
* Height and weight
* Waist circumference measurement
* Concomitant medication review
* Adverse event recording
* Urine pregnancy test
* Fasting blood assessments, e.g. hemoglobin, glucose, insulin, C-peptide, serum total and free IGF-I, IGFBP-3, C-reactive protein, adiponectin, ghrelin, non-esterified fatty acids (NEFAs), testosterone, albumin, sex hormone binding globulin and androstenedione
* Treatment exchanged to Placebo or GH

  * Visit 4, Final Assessment for the Second Treatment Phase (Week 28 +/- 1 week) (as inpatient)

The following is a description of the assessments that will be performed at the end of the second treatment phase with either GH or Placebo. Subjects will also be monitored for safety with the collection of the following:

* Physical exam and medical history
* Vital signs, e.g. pulse and blood pressure measurements
* Height and weight
* Waist circumference measurement
* Concomitant medication review
* Adverse event recording
* Urine pregnancy test
* Fasting blood assessments, e.g., hemoglobin, glucose, insulin, C-peptide, serum total and free IGF-I, IGFBP-3, C-reactive protein, adiponectin, ghrelin, non-esterified fatty acids (NEFAs), testosterone, albumin, sex hormone binding globulin and androstenedione
* A 3-hour one-step hyperinsulinemic euglycemic clamp
* MRS and DEXA scans
* Cortisol clearance rate assessments
* Fat biopsy

  * Because of the potentially long duration of Visits 1, 2 and 4, the studies can either be divided into two separate admissions upon prior arrangement or can be done all at once with one admission, depending on the subject's wishes and schedule.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age 21 to 45 years
* Body mass index between 30 to 40 kg/m2
* Diagnosis of PCOS with underlying insulin resistance (assessed by HOMA at screening visit) and/or other features that characterizes the metabolic syndrome such as hypertension ( > 130/85 mmHg), abdominal obesity (waist circumference > 88 cm), and acanthosis nigricans
* Diagnosis of normal or impaired glucose tolerance (WHO criteria)
* Stable body weight for at least 6 months prior to study entry (body weight deviating +/- 5 kg from previously recorded weight > 6 months ago)
* Normal thyroid, renal and hepatic function
* Able to self administer daily GH/Placebo injections

Exclusion Criteria:

* Inability to comply with study requirements
* Body mass index < 30 kg/m2 and > 40 kg/m2 (patients with body mass index > 40 kg/m2 are excluded because they will not fit into the MRS scanner)
* Untreated hypothyroidism or hyperthyroidism
* Anemia from any cause
* Known diabetes mellitus
* Patients with an increased risk of venous thrombosis or previous history of recurrent venous thrombosis
* Patient on any insulin-sensitizers (e.g., Metformin, Rosiglitazone, Pioglitazone) within 30 days of screening assessment
* Patient on any anti-androgens (e.g., Spironolactone, Cyproterone acetate, Flutamide, Finasteride) within 30 days of screening assessment
* Patient with other concurrent illnesses
* Pregnant (positive pregnancy test) prior enrollment in the study or planning to conceive whilst participating in the study
* Emotional/social instability likely to prejudice study completion
* Previous history of known malignancy
* Recurrent or severe unexplained hypoglycemia
* Known or suspected drug/alcohol abuse
* Patient with any metals in the body
* Any other condition/s that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Changes in insulin sensitivity, and adipocyte IGF-I and insulin receptor signaling. | 24 months

SECONDARY OUTCOMES:
Changes in body composition, cortisol production rates, and muscle and liver intramyocellular content. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C. Yuen, MRCP(UK), MD, Principal Investigator — Oregon Health and Science University; David M. Cook, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Azziz R, Woods KS, Reyna R, Key TJ, Knochenhauer ES, Yildiz BO. The prevalence and features of the polycystic ovary syndrome in an unselected population. J Clin Endocrinol Metab. 2004 Jun;89(6):2745-9. doi: 10.1210/jc.2003-032046. PMID 15181052
- [Background] Carmina E, Lobo RA. Polycystic ovary syndrome (PCOS): arguably the most common endocrinopathy is associated with significant morbidity in women. J Clin Endocrinol Metab. 1999 Jun;84(6):1897-9. doi: 10.1210/jcem.84.6.5803. No abstract available. PMID 10372683
- [Background] de Boer JA, Lambalk CB, Hendriks HH, van Aken C, van der Veen EA, Schoemaker J. Growth hormone secretion is impaired but not related to insulin sensitivity in non-obese patients with polycystic ovary syndrome. Hum Reprod. 2004 Mar;19(3):504-9. doi: 10.1093/humrep/deh122. Epub 2004 Jan 29. PMID 14998943
- [Background] Van Dam EW, Roelfsema F, Helmerhorst FH, Frolich M, Meinders AE, Veldhuis JD, Pijl H. Low amplitude and disorderly spontaneous growth hormone release in obese women with or without polycystic ovary syndrome. J Clin Endocrinol Metab. 2002 Sep;87(9):4225-30. doi: 10.1210/jc.2002-012006. PMID 12213875
- [Background] Essah PA, Nestler JE. Metabolic syndrome in women with polycystic ovary syndrome. Fertil Steril. 2006 Jul;86 Suppl 1:S18-9. doi: 10.1016/j.fertnstert.2006.04.013. PMID 16798277
- [Background] Yuen K, Wareham N, Frystyk J, Hennings S, Mitchell J, Fryklund L, Dunger D. Short-term low-dose growth hormone administration in subjects with impaired glucose tolerance and the metabolic syndrome: effects on beta-cell function and post-load glucose tolerance. Eur J Endocrinol. 2004 Jul;151(1):39-45. doi: 10.1530/eje.0.1510039. PMID 15248820
- [Background] Yuen KC, Frystyk J, White DK, Twickler TB, Koppeschaar HP, Harris PE, Fryklund L, Murgatroyd PR, Dunger DB. Improvement in insulin sensitivity without concomitant changes in body composition and cardiovascular risk markers following fixed administration of a very low growth hormone (GH) dose in adults with severe GH deficiency. Clin Endocrinol (Oxf). 2005 Oct;63(4):428-36. doi: 10.1111/j.1365-2265.2005.02359.x. PMID 16181235
- [Background] Yuen K, Frystyk J, Umpleby M, Fryklund L, Dunger D. Changes in free rather than total insulin-like growth factor-I enhance insulin sensitivity and suppress endogenous peak growth hormone (GH) release following short-term low-dose GH administration in young healthy adults. J Clin Endocrinol Metab. 2004 Aug;89(8):3956-64. doi: 10.1210/jc.2004-0300. PMID 15292333